CLINICAL TRIAL: NCT06311500
Title: Sleep Health Enhancement in Midlife Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00151143
Record Dates: First submitted 2024-01-12; First posted 2024-03-15 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Sleep Health; Midlife Adults

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep Health Enhancement Intervention (Experimental): 4 weekly visits using Zoom video conferencing consisting of education and strategies to enhance sleep health with each visit lasting about 60 minutes.
  Interventions: Behavioral: Sleep health enhancement intervention
- Wait-List Control Group (No Intervention): People in the wait-list group will continue with their usual activities for 4 weeks and then start the sleep health enhancement intervention.

INTERVENTIONS:
Behavioral: Sleep health enhancement intervention — 4 weekly visits of education and strategies to enhance sleep health
  Arms: Sleep Health Enhancement Intervention

SUMMARY:
Despite the strong links between sleep and AD, a sleep health enhancement has yet to be targeted in mid-life adults (45-64 years old) to delay or prevent AD. An intervention aimed at enhancing sleep health is a critical opportunity for primary prevention to potentially delay the onset of AD. The objective of the proposed study is to develop and assess the feasibility, acceptability, and treatment effect of a comprehensive sleep health intervention (SHI) on improving sleep health in mid-life adults

ELIGIBILITY:
Inclusion Criteria:

* 45-64 years old
* ≤ 7 on the RU-SATED self-report questionnaire
* MMSE ≥25 and AD8 <3

Exclusion Criteria:

* Known untreated sleep disorder (such as sleep apnea or restless leg syndrome)
* >3 on the STOP BANG indicating increased risk of sleep apnea
* Increased risk of restless legs syndrome on RLS-Diagnosis Index
* Evidence of circadian rhythm sleep-wake disorder
* Evidence of parasomnia
* Regular use (>2x/week) of prescription or over-the-counter medications to improve sleep
* Score of ≥15 on the Patient Health Questionnaire (PHQ-9) indicating severe depression or endorsement of any suicidal ideation (answer 1, 2 or 3 on #9 of the PHQ-9)
* Score of ≥10 on the Generalized Anxiety Disorder (GAD-7) indicating moderate to severe anxiety
* Self-report of current or history (up to 2 years) of drug or alcohol abuse based on the DSM-5-TR criteria
* History of nervous system disorder such as stroke or Parkinson's disease
* Severe mental illness such as schizophrenia or bipolar disorder
* Current or history (within 5 years) of shift work including hours of midnight-4am
* Is currently receiving a behavioral sleep health intervention

Ages: 45 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-02-13 (Actual); Primary Completion 2025-11-19 (Actual); Study Completion 2025-11-19 (Actual)

PRIMARY OUTCOMES:
6-item Acceptability Scale | immediately post-intervention
  5-point Likert scales on ease of use, understandability, enjoyment, perceived helpfulness, time commitment, and overall satisfaction
Qualitative interview | immediately post-intervention
  semi-structured interview to assess acceptability
Ru-SATED Composite score | baseline, Week 6, Week 12
  Comprised of 6 subscores (regularity, timing, efficiency, and duration from actigraphy, satisfaction from sleep diary, and alertness from Epworth Sleepiness Scale)
Sleep Self-Efficacy Scale | baseline, Week 6, Week 12
  9 item self-report Likert-scale questionnaire use to identify sleep self-efficacy.
Pittsburgh Sleep Quality Index | baseline, Week 6, Week 12
  used to assess quality of sleep
Epworth Sleepiness Scale | baseline, Week 6, Week 12
  used to assess daytime sleepiness
Dysfunctional Beliefs About Sleep (DBAS-10) consists of 10 statements reflecting beliefs and attitudes about sleep. Each statement is rated from 1 = strongly disagree to 10 = strongly agree | baseline, Week 6, Week 12
  The DBAS-10 used to identify dysfunctional beliefs about sleep
Positive Affect and Negative Affect Schedule | baseline, Week 6, Week 12
  20-item self-report questionnaire used to measure positive and negative emotions
Continuous Performance Test | baseline, Week 6, Week 12
  requires participants to respond as quickly and accurately as possible to a series of stimuli that are delivered via computer. The participants will be instructed to tap the space bar for every letter except "X."
Stroop Test | baseline, Week 6, Week 12
  requires participants to inhibit the natural response (reading a word) and replace it with another response (saying a color)
Cognitive Failures Questionnaire | baseline, Week 6, Week 12
  assesses perception of cognitive abilities over the past 6 months
Actigraphy | baseline, Week 6, Week 12
  Participants will wear an actigraph on their non-dominant wrist for 7 nights to assess sleep/wake cycle. Mains variables of interest are sleep regularity, timing, efficiency, and duration.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No